CLINICAL TRIAL: NCT05601414
Title: Cuff-less Wearable Blood Pressure Monitoring Device Validation
Brief Title: Blood Pressure Monitoring in Hypertensive Populations: Device Testing, Feasibility, Acceptability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000032876
Record Dates: First submitted 2022-10-26; First posted 2022-11-01 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Each visit will take at most 2 hours to complete study exercises. 15 Participants will have the option to complete study procedures twice more, spaced one week apart, for a total of three weeks of participation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BIO-Z vs. Finapres Nova (Experimental): Participants will have blood pressure in both arms measured three times using standard methods. The investigators will then fit the Bio-Z watch onto the non-dominant hand's wrist and the Finapres Nova® on the middle finger of the arm with the Bio-Z device. Participants will be asked to perform different exercises and blood pressure readings will be recorded during the exercise and recovery. Each exercise will be repeated three times. 15 Participants will have the option to complete study procedures twice more, spaced one week apart, for a total of three weeks of participation. Each visit will take at most 2 hours to complete study exercises for a total of 6 hours of study time if all the three visits are completed.
  Interventions: Device: BIO-Z; Device: Finapres Nova

INTERVENTIONS:
Device: BIO-Z — a novel cuffless continuous BP wrist monitor
Device: Finapres Nova — a cuffless continuous BP monitor

SUMMARY:
The goal of this study is to test a novel cuffless blood pressure (BP) monitoring device (BIO-Z) within adults with hypertension (high blood pressure) for clinical use.

The main questions it aims to answer are:

* To validate a novel cuffless blood pressure (BP) monitoring device (BIO-Z) within adults with hypertension (high blood pressure)
* To assess BP monitoring accuracy, against reference BP measurements captured by a Finapres Nova® continuous BP monitoring device in correspondence with blood pressure monitoring devices standards.

Researchers will test the device against the Finapres Nova® blood pressure monitoring device.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate a novel cuffless blood pressure monitoring device for clinical use. This device is a cuffless blood pressure watch worn on the wrist called BIO-Z. The device will be tested against the Finapres Nova® which is FDA-approved to capture continuous BP measurements. The participant will only need wear a wristband, potentially eliminating the need to perform cuff-based readings. During the 2-hour visit, research coordinators will conduct exercises to change BP and compare the values gathered by the BIO-Z watch with the Finapres Nova® device and a standard blood pressure cuff. The investigators will also test whether the Bio-Z can capture blood pressures that are in the low and high range, and whether motion affects the quality of measurement. The ultimate goal is to develop a device that passively collects blood pressure continuously, which is more convenient than a standard blood pressure cuff. 15 Participants will have the option to complete study procedures twice more, spaced one week apart, for a total of three weeks of participation.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive volunteers who have a history of hypertension or a BP >140/90 mmHg on two consecutive ambulatory visits within the last year.
* Able to read, understand, and provide written informed consent in English
* Willing and able to participate in the study procedures as described in the consent form
* Able to communicate effectively with and follow instructions from the study staff

Exclusion Criteria:

* Persons with pacemakers and/or a non-sinus rhythm (A-fib)
* Persons who are taking 4 or more anti-hypertensive medications
* Persons on dialysis
* Persons who are unstable
* Persons with tremors
* Persons with known peripheral artery disease
* Persons with more than 10 mmHg differential blood pressure between right and left arm
* Persons taking medications that might affect the hypothalamic-pituitary-adrenal axis
* The investigators will exclude persons who are known to be pregnant after 20 weeks because of physiological changes in BP after 20 weeks of pregnancy; and will refer to Electronic Health Record data to determine pregnancy status at the time of screening. The investigators will not exclude participants of childbearing age or who become pregnant during the study since there are no risk of the devices to a pregnant person.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Mean absolute difference (MAD) value between Bio-Z wristband and Finapres Nova®. | during intervention, up to 2 hours
  MAD value between the BIO-Z BP readings and the FDA- approved Finapres Nova® readings collected during the study visit will be calculated.
Mean absolute difference (MAD) value between Bio-Z wristband and Finapres Nova®. | up to 3 weeks
  MAD value between the BIO-Z BP readings and the FDA- approved Finapres Nova® readings collected during the study visit will be calculated from the sub set of 15 participants.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Spatz, Principal Investigator — Yale University
Locations (1):
- CSRU, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No